CLINICAL TRIAL: NCT03684408
Title: Use of a Radiofrequency Chip for Localization of Non-Palpable Breast Lesions: A Comparison to Wire Localization
Brief Title: Radiofrequency Chip for Localization of Non-Palpable Breast Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Health Beacons (Industry)
Responsible Party: Principal Investigator, Megha Garg, Associate Professor of Clinical Radiology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011684
Record Dates: First submitted 2018-07-27; First posted 2018-09-25 (Actual); Results first posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Breast Tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — Radio Frequency Identification Device

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- RFID and Wire Localization (Other): Part A of this project is for physician training to master the technique of RFID placement and retrieval. On the day of surgery prior to going to the operating room, all participants will have the RFID placed first to allow radiologists to become familiar with placement of the RFID localizer. Participants will then immediately undergo wire localization. Either ultrasound or mammogram guidance will be used for the localization at the discretion of the performing radiologist. Surgeons will use a reader to locate the RFID chip during surgery. The wire will be present in the event the area of concern cannot be adequately located with the reader.
  Interventions: Device: RFID and Wire Localization
- RFID Localization (Experimental): Participants will be stratified based on technique of localization (either US guidance or mammographic guidance). They will then be randomized to receive either the wire or RFID localization. There will be four visits: one pre-op breast surgery visit in which enrollment will occur, one radiology procedure visit for localization, one surgical visit, and one post-operative visit. This is the same number of visits as standard of care.
  Interventions: Device: RFID Localization
- Wire Localization (Active Comparator): Participants will be stratified based on technique of localization (either US guidance or mammographic guidance). They will then be randomized to receive either the wire or RFID localization. There will be four visits: one pre-op breast surgery visit in which enrollment will occur, one radiology procedure visit for localization, one surgical visit, and one post-operative visit. This is the same number of visits as standard of care.
  Interventions: Device: Wire Localization

INTERVENTIONS:
Device: RFID Localization — The RFID and wire localization devices used in this study are FDA approved for the image guided localization of breast tumors prior to surgical excision. The two techniques for localization will be compared in this trial.
  Arms: RFID Localization
Device: Wire Localization — The RFID and wire localization devices used in this study are FDA approved for the image guided localization of breast tumors prior to surgical excision. The two techniques for localization will be compared in this trial.
  Arms: Wire Localization
Device: RFID and Wire Localization — Both RFID and the standard of care wire localization will be performed for physician training.
  Arms: RFID and Wire Localization

SUMMARY:
The purpose of the project is to compare Radiofrequency identification device (RFID) localization technique with the current clinical standard wire localization technique. The Investigator's hypotheses is that the RFID localization technique is non-inferior to wire localization for breast lesions (tumors).

The study will be conducted in two parts. The purpose of Part A is for physician training with the RFID device. Nine subjects will undergo RFID and wire localization prior to breast lesion excision. This will allow the breast radiologists and surgeons to become comfortable with RFID device placement and retrieval. Additionally, the investigators will pilot the data collection surveys and chart review methodology to be used in Part B.

The purpose of Part B is to conduct a randomized clinical trial to assess whether RFID localization is non-inferior to wire localization for breast lesions. For this part, sixty subjects will be randomized to RFID (N=30) or wire localization (N=30) at time of enrollment. Surveys will be used to gather data from participants, radiologists, surgeons, and technologists/mammography nurses. A variety of data will be collected including, but not limited to, information on tumor size, location, depth; subject demographics; adequacy of tumor margins, re-excision rates, accuracy of wire or chip placement, and surgical complications.

DETAILED DESCRIPTION:
As part of standard of care, participants will receive: an ultrasound (US) or mammographic guided localization; excisional breast surgery; and a follow-up visit in breast surgery clinic.

As part of the research protocol, participants will receive a RFID chip for the localization procedure and complete surveys.

Part A of this project is for physician training to master the technique of RFID placement and retrieval. On the day of surgery prior to going to the operating room, all participants will have the RFID placed first to allow radiologists to become familiar with placement of the RFID localizer. Participants will then immediately undergo wire localization. Either ultrasound or mammogram guidance will be used for the localization at the discretion of the performing radiologist. Surgeons will use a reader to locate the RFID chip during surgery. The wire will be present in the event the area of concern cannot be adequately located with the reader. Participants, radiologists, surgeons, breast surgery and radiology staff will complete surveys.

Part B of this project is a prospective trial to examine safety, efficacy, operating room utilization patterns, and satisfaction with RFID versus wire localization. Participants will be stratified based on technique of localization (either US guidance or mammographic guidance). Participants will then be randomized to receive either the wire or RFID localization. There will be four visits: one pre-op breast surgery visit in which enrollment will occur, one radiology procedure visit for localization, one surgical visit, and one post-operative visit. This is the same number of visits as standard of care. Participants, radiologists, surgeons, breast surgery and radiology staff will complete surveys.

ELIGIBILITY:
Inclusion Criteria:

* Women requiring image guided pre-operative breast tumor localization

Exclusion Criteria:

* Tumors deeper than 6 cm from the skin surface
* More than one tumor requiring localization
* Tumors requiring bracketing
* Tumors requiring Magnetic Resonance Imaging localization
* Inability to complete survey
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megha Garg, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dauphine C, Reicher JJ, Reicher MA, Gondusky C, Khalkhali I, Kim M. A prospective clinical study to evaluate the safety and performance of wireless localization of nonpalpable breast lesions using radiofrequency identification technology. AJR Am J Roentgenol. 2015 Jun;204(6):W720-3. doi: 10.2214/AJR.14.13201. PMID 26001262
- [Background] Reicher JJ, Reicher MA, Thomas M, Petcavich R. Radiofrequency identification tags for preoperative tumor localization: proof of concept. AJR Am J Roentgenol. 2008 Nov;191(5):1359-65. doi: 10.2214/AJR.08.1023. PMID 18941069

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RFID and Wire Localization | RFID Localization | Wire Localization
Started | 10 | 16 | 12
Completed | 9 | 15 | 12
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RFID and Wire Localization | RFID Localization | Wire Localization | Total
Number analyzed (Participants) | 9 | 15 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 7 | 26
  >=65 years | 2 | 3 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 12 | 36
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 9 | 14 | 12 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Localization
Description: Whether the surgeon was able to identify and remove the tumor
Time Frame: From the date of localization through the date of surgery up to 4 weeks; data collected during Visit 3 at time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | RFID and Wire Localization | RFID Localization | Wire Localization
Number analyzed (Participants) | 9 | 15 | 12
Participants | 9 | 15 | 12

2. Secondary Outcome: Surveys of Satisfaction: Participant
Description: Survey Question: "Compared to expected, how uncomfortable was the localization?"
  Scored on a scale of 1 to 5 with the best being 5
Time Frame: Data collected during date of localization at Visit 2, up to approximately one month from baseline visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RFID and Wire Localization | RFID Localization | Wire Localization
Number analyzed (Participants) | 9 | 15 | 12
score on a scale | 3.4 (0.72) | 3.7 (0.85) | 4.4 (0.81)

3. Secondary Outcome: Surveys of Satisfaction
Description: Surveys of Radiology Nurse ease of scheduling the localization procedure.
  Scored on a scale of 1 to 5 with the best being 5
Time Frame: Data collected at baseline during Visit 1
Population: Not relevant for Part A. Since our breast surgeons were not experienced with using the RFID device, Part A consisted of performing the procedure with the RFID device prior to starting data collection for this outcome. This was done so that the surgeons would have completed their learning curve on a new device before data collection for this outcome began.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RFID and Wire Localization | RFID Localization | Wire Localization
Number analyzed (Participants) | 0 | 15 | 12
score on a scale |  | 4 (0.51) | 4 (1.22)

4. Secondary Outcome: Surveys of Satisfaction
Description: Surveys of radiologist satisfaction with the localization procedure.
  Scored on a scale of 1 to 5 with the best being 5
Time Frame: Data collected during date of localization at Visit 2, up to approximately one month from baseline visit
Population: Not applicable to part A. Since our breast surgeons were not experienced with using the RFID device, Part A consisted of performing the procedure with the RFID device prior to starting data collection for this outcome. This was done so that the surgeons would have completed their learning curve on a new device before data collection for this outcome began.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RFID and Wire Localization | RFID Localization | Wire Localization
Number analyzed (Participants) | 0 | 15 | 12
score on a scale |  | 4 (1.28) | 5 (1.21)

5. Secondary Outcome: Number of Participants With Tumor Incompletely Excised
Description: Number of participants with positive margin on pathology
Time Frame: Surgical resection specimen collected during Visit 3, at time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | RFID and Wire Localization | RFID Localization | Wire Localization
Number analyzed (Participants) | 9 | 15 | 12
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From localization up to surgery, up to 4 weeks, and following surgery, a maximum of 39 days
Arm/Group | RFID and Wire Localization | RFID Localization | Wire Localization
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/15 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 0/9 | 0/15 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03684408/Prot_001.pdf